CLINICAL TRIAL: NCT03912207
Title: A Human Challenge Study to Evaluate Innate and Adaptive Immune Responses to a Controlled Human Infection With BCG Administered by the Intradermal or Aerosol Inhaled Route in Healthy, BCG-naïve or Historically BCG-vaccinated, UK Adult Volunteers
Brief Title: Investigating Immune Responses to Aerosol BCG Challenge in Healthy UK Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); University of Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: TB043
Record Dates: First submitted 2019-01-30; First posted 2019-04-11 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Tuberculosis
Keywords: BCG; Aerosol; Tuberculosis; Challenge
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Volunteers in groups 1-5 will be blinded to eliminate subject bias (either conscious or subconscious) using a 10:3 randomised control design (BCG:placebo) whereby volunteers randomised to the BCG arms (Arm A) will inhale aerosolised BCG mixed with normal saline and those randomised to the placebo arms (Arm B) will inhale aerosolised normal saline.
  The volunteers will be unblinded just prior to the 3 month visit when those in Arm A may have sputum collected and those in Arm B will not. Volunteers in group 6 and 8 will not be blinded.
  For groups 1 -5, the bronchoscopist performing the procedure will also be blinded to eliminate any bias in the reporting of the appearance of the lung mucosa and extent of airway inflammation.
  All samples will be anonymised and the subject number will be allocated sequentially and therefore not identifiable with the allocated Arm. The senior immunologist will be blinded to reduce any bias that could be introduced at the sample processing stage.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Group 1, 2 Day Bronchoscopy (Experimental): Group 1: 10 volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG and 3 volunteers will receive aerosol inhaled normal saline placebo. All Group 1 volunteers will have a bronchoscopy 2 days post challenge
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 2, 7 Day Bronchoscopy (Experimental): Group 2: 10 volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG and 3 volunteers will receive aerosol inhaled normal saline placebo. All Group 2 volunteers will have a bronchoscopy 7 days post challenge
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 3, 14 Day Bronchoscopy (Experimental): Group 3: 10 volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG (Arm A) and 3 volunteers will receive aerosol inhaled normal saline placebo (Arm B). All Group 3 volunteers will have a bronchoscopy 14 days post challenge Volunteers in group 7 and group 3 (arm A) will be offered an optional follow up at 12 months, in order of enrolment until 10 such visits have been conducted. For group 3 volunteers this will be offered after unblinding.
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 4, 28 Day Bronchoscopy (Experimental): Group 4: 10 volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG and 3 volunteers will receive aerosol inhaled normal saline placebo. All Group 4 volunteers will have a bronchoscopy 28 days post challenge
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 5, 56 Day Bronchoscopy (Experimental): Group 5: 10 volunteers will receive 1 x 10^7 cfu aerosol inhaled BCG and 3 volunteers will receive aerosol inhaled normal saline placebo. All Group 5 volunteers will have a bronchoscopy 56 days post challenge
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 6, Intradermal injection, 14 Day Bronchoscopy (Experimental): Group 6: 6 volunteers will receive 1 x 10^6 cfu intradermal injection BCG + aerosol saline and will have a bronchoscopy 14 days post challenge All volunteers in group 6 will be offered an optional follow up at 12 months
  Interventions: Biological: BCG Danish; Other: Saline placebo
- Group 7, 14 Day Bronchoscopy (Experimental): Group 7: 10 volunteers will receive 1 x 10^7cfu aerosol inhaled BCG. All Group 7 volunteers will have a bronchoscopy 14 days post challenge.
  Volunteers in group 7 and group 3 (arm A) will be offered an optional follow up at 12 months, in order of enrolment until 10 such visits have been conducted
  Interventions: Biological: BCG Danish
- Group 8, Bronchoscopy Day 14 (Experimental): Group 8: 10 historically BCG vaccinated volunteers will receive aerosol inhaled BCG at a dose to be confirmed from emerging study data TB044 (Clinicaltrials.gov NCT04777721). All Group 8 volunteers will have a bronchoscopy 14 days post challenge.
  Interventions: Biological: BCG Danish

INTERVENTIONS:
Biological: BCG Danish — BCG Danish 1331 is on the WHO list of pre-qualified vaccines and has a well-defined side effect profile. BCG is licensed for delivery via the intradermal route. It is not licensed for delivery via the aerosol route.
Other: Saline placebo — Saline is a routinely used placebo.
  Arms: Group 1, 2 Day Bronchoscopy; Group 2, 7 Day Bronchoscopy; Group 3, 14 Day Bronchoscopy; Group 4, 28 Day Bronchoscopy; Group 5, 56 Day Bronchoscopy; Group 6, Intradermal injection, 14 Day Bronchoscopy

SUMMARY:
TB043 is a clinical challenge trial primarily to evaluate the safety of BCG challenge administered by the aerosol inhaled route in healthy, BCG naive (Group 1-7) as well as historically BCG vaccinated UK adults (Group 8) . The trial will also look to evaluate and compare the amount of BCG recovered from the lungs as various points after challenge.

DETAILED DESCRIPTION:
Mycobacterium tuberculosis (M.tb) is a pathogen with worldwide preponderance that infects humans and causes the transmissible disease tuberculosis (TB). An estimated one-third of the world's population is latently infected with M.tb, carrying a 10% lifetime risk of developing active life-threatening disease. In 2016, there were 10 million new cases worldwide and 1.7 million people died of TB. Co-infection with human immunodeficiency virus (HIV) greatly increases the risk of TB reactivation and death. Diagnosis is challenging and drug treatment is often harmful, costly and complex. For these reasons, it is essential to develop a more effective vaccine against TB.

An improved understanding of the nature of protective immunity in humans would significantly improve rational vaccine development. Whilst host immunity, particularly systemic adaptive immunity, has been well characterized in murine models, the understanding of the immunological events that occur in humans during acute infection is limited. In particular, the knowledge of human mucosal responses to M.tb. is limited. This is primarily due to the difficulties in studying early disease processes in the lung. Consequently, the majority of human studies have investigated immune responses ex-vivo in peripheral blood or after in-vitro infection of cell lines. A better understanding of the immune components that exist at the respiratory mucosal surfaces in humans could lead to interventions that prevent infection at the point of entry.

TB043 is a clinical challenge trial primarily to evaluate the safety of BCG challenge administered by the aerosol inhaled route in healthy, BCG naive (Group 1-7) as well as historically BCG vaccinated UK adults (Group 8) . The trial will also look to evaluate and compare the amount of BCG recovered from the lungs as various points after challenge, allowing investigation into the immune components at mucosal surfaces.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18-50 years
* Resident in or near Oxford for the duration of the study period
* Screening IGRA negative
* No relevant findings in medical history or on physical examination
* Allow the Investigators to discuss the individual's medical history with their GP
* Use effective contraception (see below) for the duration of the study period (people of child bearing potential only)
* Refrain from blood donation during the study
* Give written informed consent
* Allow the Investigator to register volunteer details with a confidential database (The Over-volunteering Protection Service) to prevent concurrent entry into clinical studies/trials
* Willing to be tested for evidence of SARS-CoV-2 infection, if indicated and to allow public health notification of results if required.
* Able and willing (in the Investigator's opinion) to comply with all the study requirements
* For Group 8 only- previously vaccinated with BCG (at least 12 months prior to enrolment, as evidenced by a visible scar or documentation in medical or occupational health records)

Exclusion Criteria:

* Previously resident for more than 12 months concurrently in a rural area of a tropical climate where significant non-tuberculous mycobacterial exposure is likely
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior vaccination with BCG (G1-7 only) or any other candidate TB vaccine (all groups).
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned study challenge date
* Clinically significant history of skin disorder, allergy, atopy, immunodeficiency (including HIV), cancer (except BCC or CIS), cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness, psychiatric disorder, drug or alcohol abuse
* Concurrent oral, inhaled or systemic steroid medication or the concurrent use of other immunosuppressive agents
* Shares a household with someone with clinically significant immunodeficiency (either from infection or medication) who is deemed to be at risk of developing disseminated BCG infection if exposed to BCG
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the study agent, essential study procedures, sedative drugs, or any local or general anaesthetic agents
* Pregnancy, lactation or intention to become pregnant during study period
* Any clinically significant respiratory disease, including asthma
* Current smoker (defined as any smoking including e-cigarettes in the last 3 months)
* Clinically significant abnormality on screening chest radiograph
* Clinically significant abnormality of pulmonary function
* Any nasal, pharyngeal, or laryngeal finding which precludes bronchoscopy
* Current use of any medication taken through the nasal or inhaled route including cocaine or other recreational drugs
* Clinical, radiological, or laboratory evidence of current active TB disease
* Past treatment for TB disease
* Any clinically significant abnormality of screening blood or urine tests
* Positive HBsAg, HCV or HIV antibodies
* Any other significant disease, disorder, or finding, which, in the opinion of the Investigator, may either put the volunteer at risk, affect the volunteer's ability to participate in the study or impair interpretation of the study data

People of Child Bearing Potential (POCBP) are required to use an effective form of contraception during the course of the study.

Acceptable forms of contraception for POCBP volunteers include:

* Established use of oral, injected on implanted hormonal methods of contraception
* Placement of an intrauterine device (IUD) or intrauterine system (IUS)
* Permanent sterilisation or bilateral tubal occlusion
* Barrier methods of contraception (condom; or occlusive cap with spermicide)
* Male sterilisation, if the vasectomised partner is the sole partner for the subject
* True abstinence, when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence and withdrawal are not acceptable methods of contraception)
* Exclusive same sex intercourse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2019-04-19 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Identification of markers of innate immunity-cytokines | Up to day 168
  Established markers of innate immunity in blood, BAL and biopsy samples will be aggregated to determine overall characterisation of innate response. Specifically, cytokine levels will be measured by ELISpot and ELISA.
Identification of markers of innate immunity-antigen presenting cells | Up to day 168
  Established markers of innate immunity in blood, BAL and biopsy samples will be aggregated to determine overall characterisation of innate response. Specifically, the activity of antigen presenting cells will be measured by flow cytometry
Identification of markers of innate immunity-inflammation in tissue | Up to day 168
  Established markers of innate immunity in blood, BAL and biopsy samples will be aggregated to determine overall characterisation of innate response. Specifically IHC staining will be done to examine changes in tissue samples.
Identification of markers of adaptive immunity-antibodies | Up to day 168
  Established markers of adaptive immunity in blood, BAL and biopsy samples will be aggregated to determine overall characterisation of adaptive response. Specifically, the presence of antibodies will be measured.
Identification of markers of adaptive immunity-T cells | Up to day 168
  Established markers of adaptive immunity in blood, BAL and biopsy samples will be aggregated to determine overall characterisation of adaptive response. Specifically, T-cell activity will be determined by a flow cytometry panel.

SECONDARY OUTCOMES:
Mycobacterial growth inhibition assay | Up to day 56
  MGIA outcome on PBMCs collected at Day 56; readout in CFUs (colony forming units)

OTHER OUTCOMES:
Adverse Events (AEs) | Up to day 168
  Collection of AE data at each visit and via diary card, and laboratory parameters of BCG cfu counts in induced sputum, BAL and matrix from adapted duck bill mask collection

CONTACTS AND LOCATIONS:
Overall Officials: Professor Helen McShane, Principal Investigator — University of Oxford
Locations (2):
- United Kingdom (2):
  - Centre for Clinical Vaccinology and Tropical Medicine (CCVTM), Churchill Hospital, Oxford, Oxfordshire
  - Oxford University Hospitals- John Warin Ward, University of Oxford, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No